CLINICAL TRIAL: NCT04155255
Title: My Body is Fit and Fabulous: an Intervention Program to Combat Obesity Among Malaysian School Children
Brief Title: My Body is Fit and Fabulous at School Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Health, Malaysia (Other Government); Ministry of Education, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRR1343916563
Record Dates: First submitted 2019-10-06; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Overweight, Childhood
MeSH Terms: conditions — Pediatric Obesity

ARMS (2):
- Control (No Intervention): Age-matched overweight and obese students were selected from control schools. The students participated in their usual health and physical education classes plus any other curriculum activities provided by the school.
- Intervention (Experimental): Overweight and obese students were recruited from intervention schools. Students underwent MyBFF@school intervention programme that consisted of physical activity, nutrition and psychological modules for the duration of 6 months. MyBFF@school intervention programme were conducted by trained personnel that were stationed full-time at each intervention school.
  Interventions: Other: MyBFF@school

INTERVENTIONS:
Other: MyBFF@school
  Arms: Intervention

SUMMARY:
"My Body is Fit and Fabulous" (MyBFF@school) program was designed specifically for overweight and obese school children in order to help them control their BMI and body fat. MyBFF@school is a multi-faceted obesity intervention program that incorporated physical activity, nutrition and psychology modules.

DETAILED DESCRIPTION:
"My Body is Fit and Fabulous" (MyBFF@school) is a school-based, cluster randomised controlled trial (C-RCT) study that primarily aimed to evaluate the effectiveness of MyBFF@school program on overweight and obese school childrens' BMI for age (BMI z-score) and body fat percentage at 3 and 6 months post intervention. Primary and secondary schools in the central region of Peninsular Malaysia were randomised to either intervention or control school via systematic random sampling method. The selected intervention schools underwent MyBFF@school programme that consisted of physical activity, nutrition and psychology modules, whereas the control schools followed the standard national school curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Give consent
* Overweight and obese students with BMI for age (BMI z-score) more than +1SD based on WHO 2007 Growth Reference
* Age between 9-16 years old

Exclusion Criteria:

* BMI for age below and equal +1SD
* Physical or mental disability
* Medical conditions that prevent him/her to participate in moderate-to-vigorous physical activity
* Co-morbidities that may interfere with the study such as:

  1. diagnosed type 2 diabetes mellitus
  2. hypertension
  3. nephritic syndrome
  4. epilepsy
  5. congenital heart disease
  6. skeletal anomalies
* On steroids
* On anti-epileptic
* On methylphenidate

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2438 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
BMI z-score | Change from Baseline BMI z-score at 3 months and change from Baseline BMI z-score at 6 months
  To see changes in BMI z-score. Also called as BMI standard deviation scores, which measures relative weight adjusted for child age and sex. Weight in kilograms and height in meters will be combined to report BMI in kg/m^2. By using the value of BMI obtained, BMI z-score was calculated using World Health Organization (WHO) AnthroPlus 2007 software, with indication of overweight >+1.0 SD, obese >+2.0 SD and morbidly obese >+3.0 SD.
Percentage of Body Fat (%) | Change from Baseline Body Fat Percentage at 3 months and change from Baseline Body Fat Percentage at 6 months
  To see changes in percentage of body fat. It is the percentage of body weight that is made up of fat. It consists of both storage body fat and essential body fat. It was measured in light clothing without shoes and socks to the nearest 0.1 kg using a pre-calibrated body impedance analyser (InBody 770, Korea)
Waist Circumference (cm) | Change from Baseline Waist Circumference at 3 months and change from Baseline Waist Circumference at 6 months
  To see changes in Waist Circumference. Waist Circumference was measured twice to the nearest 0.1 cm over the skin midway between the tenth rib and the iliac crest at the end of normal expiration, using a non-extensible tape.
Skeletal Muscle Mass (kg) | Change from Baseline Skeletal Muscle Mass at 3 months and change from Baseline Skeletal Muscle Mass at 6 months
  To see changes in Skeletal Muscle Mass. Skeletal Muscle Mass is the weight of muscles that connected to the bones in the body that were measured in light clothing without shoes and socks to the nearest 0.1 kg using a pre-calibrated body impedance analyser (InBody 770, Korea)

SECONDARY OUTCOMES:
HbA1c Level | Change from Baseline HbA1c Level at 6 months.
  To see changes in HbA1c Level. HbA1c level was determined by cationic exchanged high performance liquid chromatography (Adams A1c HA-8160, Arkray Inc, Japan) and followed the National Glycohemoglobin Standardization Programme Guidelines.
Fasting Plasma Glucose | Change from Baseline Fasting Plasma Glucose at 6 months.
  To see changes in Fasting Plasma Glucose. Fasting Plasma Glucose was analysed by Randox Laboratories (Antrim, UK) using an auto chemical analyser (Dirui CS-400, China).
Total Cholesterol | Change from Baseline Total Cholesterol at 6 months.
  To see changes in Total Cholesterol. Total Cholesterol was analysed by Randox Laboratories (Antrim, UK) using an auto chemical analyser (Dirui CS-400, China). The cut-off value for high Total Cholesterol is 5.20 mmol/L.
Triglycerides Level | Change from Baseline Triglycerides Level at 6 months.
  To see changes in Triglycerides Level. Triglycerides Level was analysed by Randox Laboratories (Antrim, UK) using an auto chemical analyser (Dirui CS-400, China). The cut-off value for high Triglycerides Level is 1.70 mmol/L.
HDL-C Level | Change from Baseline HDL-C Level at 6 months.
  To see changes in HDL-C Level. HDL-C Level was analysed by Randox Laboratories (Antrim, UK) using an auto chemical analyser (Dirui CS-400, China). The cut-off value for low HDL-C Level is 1.03 mmol/L.
LDL-C Level | Change from Baseline LDL-C Level at 6 months.
  To see changes in LDL-C Level. LDL-C Level was analysed by Randox Laboratories (Antrim, UK) using an auto chemical analyser (Dirui CS-400, China). The cut-off value for high LDL-C Level is 2.84 mmol/L.
Fasting Insulin Level | Change from Baseline Fasting Insulin Level at 6 months.
  To see changes in Fasting Insulin Level. Fasting Insulin levels were measured using an automated enzyme immunoassay analyser (TOSOH AIA-360, Japan).
HOMA-IR | Change from Baseline HOMA-IR at 6 months.
  To see changes in HOMA-IR. HOMA-IR is calculated by multiplying the value of fasting insulin and fasting plasma glucose and divided by 22.5.
TG:HDL-C Ratio | Change from Baseline TG:HDL-C Ratio at 6 months.
  To see changes in TG:HDL-C Ratio. TG:HDL-C Ratio is calculated by dividing triglycerides levels with HDL-C levels.
Physical Fitness Score | Change from Baseline Physical Fitness Score at 3 months and change from Baseline Physical Fitness Score at 6 months
  To see changes in Physical Fitness Score. Physical Fitness Score was assessed using Modified Harvard Step Test. Physical Fitness Score was calculated with this formula: (Total duration in seconds/Total pulse rate at 0, 1 and 2 minutes) X 100. After the calculation of the physical fitness score, the subjects' physical fitness were categorized into 5 different categories. The first category was poor, where the score of their physical fitness score is below 54. The second was low average, as their physical fitness score falls between the range of 55 to 64. Next, high average with the score between 65 to 79 followed by the fourth category which was good i.e. between the ranges of 80 to 89. Lastly, the fifth category was excellent, where the subjects' physical fitness score were more than 90.
Nutrition Knowledge | Change in Nutrition Knowledge from Baseline to 6 months assessment
  To assess their changes of Nutrition Knowledge using a pre-tested Nutrition Knowledge using a validated Nutrition Knowledge Questionnaire. The school children completed a 10-item True/ False/ Don't know Nutrition Knowledge questionnaire before and after intervention. The correct answer was given a score of 1 whereas for the wrong answer and I don't know was given a score of 0. The total score for every respondent was calculated from the correct responses with a maximum of 10 points which were then converted to percentages. Total scores for the knowledge items were then ranked into 3 tertiles; lowest (≤50%), middle (60%) and highest (70-100%).
Nutrition Attitude | Change in Nutrition Attitude from Baseline to 6 months assessment
  To assess their changes of Nutrition Attitude using a pre-tested Nutrition Attitude Questionnaire. There were 15 questions for the attitude items. The attitude items were on a five-point Likert scale ranging from strongly disagree (1 point) to strongly agree (5 points). An intermediate (neutral) option was allocated 3 points. Total scores for the attitude items were then ranked into 3 tertiles; lowest (≤50%), middle (60%) and highest (70-100%).
Nutrition Practice | Change in Nutrition Practice from Baseline to 6 months assessment
  To assess their changes of Nutrition Practice using a pre-tested Nutrition Practice Questionnaire. Assessment focused mainly on the key components that should be and commonly practiced by the school children. These included intake of fruit and vegetable, plain water, carbonated drinks, breakfast intake a swell as food commonly brought food from home and also food commonly purchased from the school canteen.
Stages of Change for Weight Management (Secondary School) | Change in behaviour of weight management from Baseline to 6 months assessment
  To assess their behavioural changes via Stage of Change of Weight Management by using a validated Trans Theoretical Model Questionnaire for weight management behaviour.
Stages of Change for Fruit and Vegetable Intake (Secondary School) | Change from Baseline Stages of Change of Fruit and Vegetable Intake at 6 months
  To assess their behavioural changes via Stage of Change of Fruit and Vegetable Intake by using a validated Trans Theoretical Model Questionnaire for fruit and vegetable intake behaviour.
Health-Related Quality of Life (Primary School) | Change in behaviour of fruit and vegetable intake from Baseline to 6 months assessment
  To assess their changes of Health-Related Quality of Life using KINDL-R questionnaire. It contains 24 Likert-scaled items that are associated with 6 subscales namely physical well-being, emotional well-being, self-esteem, friend, family and school functioning. Total scores are obtained by adding the scores of all subscales. Higher scores represent better outcome. Range score from 15 to 75
Well-Being (Primary School) | Change from Baseline Well-Being at 6 months
  To assess their changes of Well-Being using the Stirling Children Well-being Scale (SCWBS) questionnaire. It is comprised of two subscales which are positive outlook and positive emotional state. Total scores are obtained by adding the scores of all subscales. Higher scores represent better outcome. Range score from 24 to 120
Eating Attitude (Primary School) | Change from Baseline Eating Attitude at 6 months
  To assess their changes of Eating Attitude using the Children' Eating Attitude Test (ChEAT) questionnaire. It is comprised of three subscales namely dieting, restricting and purging, food and oral control . Higher scores represent worse outcome. Range score from 26 to 156
Emotional and Psychological Well-Being (Secondary School) | Change from Baseline Emotional and Psychological Well-Being at 6 months
  To assess their changes of Emotional and Psychological Well-Being using the Youth-Self Report questionnaire. YSR contains 112 items to measure emotional and behavioral problems comprising of 12 subscales which are anxious /depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behaviour, aggressive behaviour, other problems, internalizing, externalizing and total behaviour. Internalizing are the total sum of the subscales of anxious/depressed, withdrawn/depressed and somatic complaints. Externalizing are the total sum of rule-breaking behaviour and aggressive behaviour. Total behavior are the sume of all subscales. Higher scores represent worse outcome. Range score from 0 to 224
Eating Attitude (Secondary School) | Change from Baseline Eating Attitude at 6 months
  To assess their changes of Eating Attitude using the Eating Attitude Test (EAT-26) questionnaire. It is comprised of three subscales namely dieting, bulimia and food preoccupation and oral control. Higher scores represent worse outcome. Range score from 30 to 180
Healthy Eating Behavior (Secondary School) | Change from Baseline Healthy Eating Behavior at 6 months
  To assess their changes of Healthy Eating Behavior using the Adolescents Food Habits Checklist. Higher scores represent better outcome. Range score from 0 to 46

OTHER OUTCOMES:
Blood Pressure | Change from Baseline Blood Pressure at 6 months.
  To see changes in Blood Pressure. Blood Pressure reading was measured manually by trained staffs using a mercury sphygmomanometer (Accoson, UK) with appropriate cuff size for each individual.
Baseline Pubertal Status | Baseline
  Pubertal Status was assessed (self-administered) using Tanner staging scale.
Pubertal Status Post-Intervention | At 6 months
  Pubertal Status was assessed (self-administered) using Tanner staging scale.
Acanthosis Nigricans | Baseline
  Participants were examined for the presence of acanthosis nigricans over the neck.

REFERENCES:
- [Derived] Ishak Z, Fin LS, Ibrahim WAHW, Yahya A, Zain FM, Selamat R, Jalaludin MY, Mokhtar AH. The effectivess of MyBFF@school intervention program in reducing emotional and behavioral problems in overweight and obese secondary schoolchildren in Malaysia: a cluster randomized controlled trial. BMC Public Health. 2025 Jul 28;24(Suppl 1):3631. doi: 10.1186/s12889-025-23545-y. PMID 40721745
- [Derived] Jalaludin MY, Zin RMWM, Roslan FA, Mansor F, Zain FM, Hong JYH, Kamil NZIA, Yahya A, Ishak Z, Selamat R, Mokhtar AH. Cardiometabolic outcome of MyBFF@school intervention program among primary schoolchildren: a cluster randomized controlled trial. BMC Public Health. 2025 Jul 24;24(Suppl 1):3630. doi: 10.1186/s12889-025-23546-x. PMID 40702531
- [Derived] Selamat R, Aziz NAA, Raib J, Zulkafly N, Mohamad WAW, Ismail AN, Jalaludin MY, Zain FM, Ishak Z, Yahya A, Mokhtar AH. Effects of a nutrition education intervention on nutrition knowledge and attitude among overweight and obese primary schoolchildren: a cluster randomized controlled trial. BMC Public Health. 2025 Feb 4;24(Suppl 1):3629. doi: 10.1186/s12889-025-21671-1. PMID 39905418
- [Derived] Zin RMWM, Mokhtar AH, Yahya A, Zain FM, Selamat R, Ishak Z, Jalaludin MY. Effects of MyBFF@school, a multifaceted obesity intervention program, on anthropometry and body composition of overweight and obese primary schoolchildren. BMC Public Health. 2025 Jan 14;24(Suppl 1):3627. doi: 10.1186/s12889-024-20724-1. PMID 39810108
- [Derived] Mokhtar AH, Zin RMWM, Yahya A, Zain FM, Selamat R, Ishak Z, Jalaludin MY. Rationale, design, and methodology of My Body Is Fit and Fabulous at school (MyBFF@school) study: a multi-pronged intervention program to combat obesity among Malaysian schoolchildren. BMC Public Health. 2025 Jan 10;24(Suppl 1):3626. doi: 10.1186/s12889-024-20726-z. PMID 39794750
- [Derived] Selamat R, Raib J, Aziz NAA, Zulkafly N, Ismail AN, Mohamad WNAW, Zulkiply AA, Jalaludin MY, Zain FM, Ishak Z, Yahya A, Mokhtar AH. Effects of the MyBFF@school obesity intervention program with nutrition education intervention on nutrition knowledge and attitude of secondary schoolchildren: a cluster randomized controlled trial. BMC Public Health. 2025 Jan 9;24(Suppl 1):3624. doi: 10.1186/s12889-024-21090-8. PMID 39789494
- [Derived] Kamil NZIA, Mokhtar AH, Yahya A, Zain FM, Selamat R, Ishak Z, Jalaludin MY. Effects of the MyBFF@school program on anthropometry and body composition among overweight and obese adolescent schoolchildren. BMC Public Health. 2025 Jan 9;24(Suppl 1):3625. doi: 10.1186/s12889-024-20725-0. PMID 39789486
- [Derived] Mokhtar AH, Kamarudin MA, Choong A, Singh L, Genisan V, Yahya A, Zin RMWM, Zain FM, Selamat R, Ishak Z, Jalaludin MY. The effect of the MyBFF@school program on cardiorespiratory fitness in overweight and obese primary schoolchildren: a cluster randomized controlled trial. BMC Public Health. 2025 Jan 9;24(Suppl 1):3623. doi: 10.1186/s12889-024-20723-2. PMID 39789464